CLINICAL TRIAL: NCT01798771
Title: Intraoperative MRI and 5-ALA Guidance to Improve the Extent of Resection in Brain Tumor Surgery
Acronym: IMAGER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Christian Senft, PD Dr. med. Christian Senft, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JohannWGUH_IMAGER; 206/12 (Other: Ethics Committee Johann Wolfgang Goethe University)
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Primary Malignant Neoplasm of Nervous System; Glioma; Glioblastoma; Metastasis
Keywords: primary brain tumor; malignant glioma; intraoperative MRI; 5-ALA
MeSH Terms: conditions — Glioma; Glioblastoma; Neoplasm Metastasis; Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Control arm (Other): 5-ALA fluorescence guided surgery in patients with contrast enhancing tumors.
  Interventions: Procedure: Control arm
- Interventional arm (Other): 5-ALA fluorescence guided surgery with the additional use of an intraoperative MRI for resection control in patients with contrast enhancing tumors.
  Interventions: Procedure: Interventional arm

INTERVENTIONS:
Procedure: Interventional arm — 5-ALA fluorescence guided surgery with the additional use of an intraoperative MRI for resection control in patients with contrast enhancing tumors.
  Other Names: 5-ALA; 5-Aminolevulinic acid hydrochloride
  Arms: Interventional arm
Procedure: Control arm — 5-ALA fluorescence guided surgery in patients with contrast enhancing tumors.
  Other Names: 5-ALA; 5-Aminolevulinic acid hydrochloride
  Arms: Control arm

SUMMARY:
The investigators hypothesize that the rate of radiologically complete resections of contrast-enhancing brain tumors following surgeries aided by use of 5-ALA induced fluorescence guidance and use of an intraoperative ultra-low field MRI is higher compared to surgeries aided by 5-ALA induced fluorescene alone.

ELIGIBILITY:
Inclusion Criteria:

* adult patient (> 18 years) able to give informed consent
* primary supratentorial intra-axial brain tumor exhibiting contrast enhancement suspected to be malignant glioma
* tumor must be deemed completely resectable by neurosurgeon
* diagnostic MRI

Exclusion Criteria:

* patient unable or unwilling to give informed consent
* infratentorial tumor location
* tumor location in or near eloquent areas
* multifocal tumor
* existance of contraindications to undergo MRI examination
* previous surgical treatment for an intraaxial brain tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Extent of Resection | Early postoperative MRI within 72 hrs
  The primary efficacy endpoint is the rate of complete resections according to early postoperative MRI.

SECONDARY OUTCOMES:
Volumetric extent of resection | Early postoperative MRI within 72hrs
  Secondary endpoint is the volumetric extent of resection as determined by direct comparison of preoperative and early postoperative tumor volumes.
PFS 6 | 6 months following surgery
  Secondary endpoint is the rate of subjects with progression-free survival (PFS) 6 months after tumor resection
PFS 12 | 12 months following surgery
  Secondary endpoint is the rate of subjects with progression-free survival (PFS) 12 months after tumor resection
Quality of life | 6 months/12 months
  Patient quality of life at 6 and 12 months following surgery is a secondary endpoint

OTHER OUTCOMES:
NIHSS | 5 days following surgery
  The change of NIHSS (The NIH Stroke Scale) score is an other pre-specified outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Christian Senft, MD PhD, Principal Investigator — Dept. of Neurosurgery, Johann Wolfgang Goethe University Hospital
Locations (1):
- Klinik für Neurochirurgie Johann Wolfgang Goethe University, Frankfurt am Main, Hesse, Germany